CLINICAL TRIAL: NCT06722430
Title: A Phase 1 Open-label Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of Icalcaprant in Healthy Adult Subjects
Brief Title: A Study to Assess Change in How Oral Icalcaprant With Itraconazole Moves Through the Body in Healthy Adult Participants
Acronym: 529 DDI ITZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M25-529
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Icalcaprant; Itraconazole; ABBV-1354; CVL-354
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Icalcaprant with Itraconazole (Experimental): Participants will receive oral Icalcaprant with Itraconazole up to 8 days and then followed for 30 days.
  Interventions: Drug: Icalcaprant; Drug: Itraconazole (ITZ)

INTERVENTIONS:
Drug: Icalcaprant — Oral capsule
  Other Names: ABBV-1354; CVL-354
Drug: Itraconazole (ITZ) — Oral capsule

SUMMARY:
This study is to assess the change of itraconazole, a strong CYP3A inhibitor, on the pharmacokinetics, safety, and tolerability of a single dose of icalcaprant in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of any clinically significant sensitivity or allergy to any medication or food.
* Exposure to icalcaprant within the past 90 days.
* History of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption [e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, gastric surgery (except pyloromyotomy for pyloric stenosis during infancy), cholecystectomy, vagotomy, bowel resection, etc.].

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Icalcaprant | Up to approximately 14 days
  Cmax of Icalcaprant
Time to Cmax (Tmax) of Icalcaprant | Up to approximately 14 days
  Tmax of Icalcaprant
Terminal Phase Elimination Rate Constant (Beta) of Icalcaprant | Up to approximately 14 days
  Beta of Icalcaprant
Terminal Phase Elimination Half-Life (t1/2) of Icalcaprant | Up to approximately 14 days
  T1/2 of Icalcaprant
Area under the plasma concentration-time curve (AUC) of Icalcaprant | Up to approximately 14 days
  AUC of Icalcaprant
Area under the plasma concentration-time curve from time 0 until the last measurable Concentration (AUCt) of Icalcaprant | Up to approximately 14 days
  AUCt of Icalcaprant
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) of Icalcaprant | Up to approximately 14 days
  AUCinf of Icalcaprant
Number of Participants with Adverse Events (AEs) | Up to approximately 47 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 271617, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-529